CLINICAL TRIAL: NCT03208348
Title: Low-Cost, Virtual Reality System to Increase Access to Exposure Therapy for Anxiety and Obsessive Compulsive Disorders
Brief Title: Pilot Study of Virtual Reality for Providing Exposure Therapy to Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota HealthSolutions (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Virtual Reality
Record Dates: First submitted 2017-06-01; First posted 2017-07-05 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: A single group will pilot test a virtual reality system that is designed to support mental health treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot virtual reality (Experimental): Children with anxiety will have a single visit to test the virtual reality system and measure its affects on their anxiety ratings.
  Interventions: Other: Pilot Virtual Reality

INTERVENTIONS:
Other: Pilot Virtual Reality — Exposure to a virtual reality vignette with anxiety rating to support exposure therapy

SUMMARY:
Drs. from the Mayo Clinic Rochester will plan and execute a feasibility study of the phase I prototype version of the Virtual Reality exposure therapy system. Dr. X, who has significant experience in evaluating patient experiences and opinions of technologies intended to change behavior, will oversee a qualitative study to examine the prototype system. Twenty children with generalized anxiety disorder with perfectionism who have received less than 3 treatment sessions and a parent will be recruited to pilot the Virtual Reality system.

DETAILED DESCRIPTION:
Twenty children with generalized anxiety disorder (perfectionism) who have received less than 3 treatment sessions and a parent will be recruited to pilot the Virtual Reality system. Participants will be identified through the Mayo Clinic Pediatric Anxiety Disorders Clinic (PADC) using purposive sampling methods. Each patient will participate in a single (up to) 2-hour visit, allowing for breaks as needed. Staff from Mayo Clinic HealthCare Policy & Research experienced in qualitative data analysis and not involved with the patients' medical care or development of the prototype system will conduct the study visits. During the first 30 minutes the patient and parent will be introduced to the Virtual Reality system and the rationale for this feasibility study. Next, a therapist from the PADC, all of whom are experienced exposure therapists, will lead the patient through exposure exercises using the Virtual Reality system for up to 30 minutes. During the next period, up to 30 minutes, the therapist will go to a different room and the patient, with support from their parent, will complete exposure exercises using the Virtual Reality system that the therapist directed them to complete. During the exposures the interviewer will observe, code and record the patient's interaction with the Virtual Reality system. The data from the Virtual Reality system will be automatically transmitted to a cloud service running on a local laptop to study the effectiveness of the system's automatic logging capabilities. For the remaining time (up to 30 minutes) the interviewer will interview the patient about his or her experience with the Virtual Reality system and then will ask for observations and opinions from the parent.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Generalized Anxiety Disorder with perfectionism and have received less than three treatment sessions

Exclusion Criteria:

* too young to safely and effectively participate with the study materials

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Qualitative response to the system as assessed by observation while using the system and interview following use. | through study completion, an average of one day study visit
  Twenty participants will provide qualitative data about their experience using the system.

SECONDARY OUTCOMES:
Anxiety as assessed by the Subjective Units of Distress Scale | through study completion, an average of one day study visit
  Anxiety for each of the twenty participants will be assessed using SUDS prior to and after each time repeating the exposure. Participants will self-select how many times to repeat the exposure during the one day study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Seifert, MPH, Principal Investigator — Minnesota HealthSolutions
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No